CLINICAL TRIAL: NCT03203122
Title: The Effect of Intense Pulsed Light Assisted Hair Removal Therapy on Mild and Moderate Cases of Hidrosadenitis Suppurativa
Brief Title: Intense Pulsed Light Therapy for Hidrosadenitis Suppurativa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REG-115-2016
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Hidradenitis Suppurativa; Acne Inversa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: Patients are randomized to treatment in either left or right side, using the other side as control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assesor and primary invstigator are blinded and not present at treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients are randomized to treatment of either right or left side. The other side works as control
  Interventions: Other: IPL laser
- Comparator Group (Sham Comparator): Patients are randomized to treatment in either right or left side. The other side works as control
  Interventions: Other: No sham treatment

INTERVENTIONS:
Other: IPL laser — IPL laser monthly. Vertical and horizontal treatment, one pass over. Settings according to fitzpatrick skin type
  Arms: Study group
Other: No sham treatment — The treatment is slightly painful, and noisy. Sham treatment impossible
  Arms: Comparator Group

SUMMARY:
6 monthly treatments with IPL laser in patients with Hidradenitis Suppurativa. The effect in measured on several severity scores.

DETAILED DESCRIPTION:
Patient suffering from bilateral HS in the axilla or groin area are threated with IPL laser monthly for 6 months.

Patients are randomized to treatment in either left or right side, the other side works as control.

No sham treatment, but observers are blinded.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral HS in the axilla or groin area
* Fitzpatrick skin type I-II

Exclusion Criteria:

* Pregnant
* Unable to understand or communicate with study personnel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-07 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
HiScore | After 6 treatments i.e. 6 months
  50 % reduction in abcesses and draining fistual

SECONDARY OUTCOMES:
Sartorius score | after 6 treatments i.e. 6 months
  HS severity score
Physician global assesment | after 6 treatments i.e. 6 months
  HS severity score

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Zealland, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No
Will not be shared